CLINICAL TRIAL: NCT04025749
Title: Executive Training in Cerebral Palsy: Participation, Quality of Life and Brain Connectivity
Brief Title: Cognitive Training Cerebral Palsy
Acronym: ETCONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Generalitat de Catalunya (Unknown)
Responsible Party: Principal Investigator, Roser Pueyo, Associate professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSI2016-75979-R AEI/FEDER, UE; 2017SGR748 (Other Grant/Funding Number: Generalitat de Catalunya)
Record Dates: First submitted 2019-06-11; First posted 2019-07-19 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Executive Functions; Cognitive Training; Computerized Therapy; Quality of Life; Neuroimaging; Participation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention group (Experimental): Thirty children with CP aged 8 to 12 years (or fifteen with neuroimage data) will participate in a computerized executive training program from home (12 weeks, 5 days a week, 30 min a day).
  Interventions: Behavioral: Computerized Executive Functions training
- Wait-list delayed intervention (Other): Thirty children with CP (or fifteen with neuroimage data) matched by age, sex, motor and cognitive impairment severity.
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: Computerized Executive Functions training — Home-based executive function training with adaptive difficulty, through NeuronUp (https://www.neuronup.com) over 12 weeks (30 min/day, 5 days per week, 30h in total).
  Arms: Immediate intervention group
Other: Care as usual — Care as usual
  Arms: Wait-list delayed intervention

SUMMARY:
This study aims to conduct a single-blind randomized controlled trial with sixty children with Cerebral Palsy (CP) to explore if a home-based computerized multi-modal executive training is effective improving infants' executive functions (EF), as the primary outcome. As secondary outcomes, it will be tested if the intervention exerts a positive effect on other cognitive functions, social relationships, and quality of life (QOL) in children with CP. It is expected to observe changes in brain structure and functioning associated to clinical improvements.

The primary hypothesis to be tested is that a computerized multi-modal cognitive training will be more effective at improving EF than usual care alone.

Secondary hypotheses are that the computerized therapy will be more effective than usual care alone at improving specific cognitive functions such as visuoperception, memory, social relationships and QOL. In addition, we also hypothesize there will be changes on brain structure and function. We further hypothesise that these changes will be maintained over time (9 months). Finally, sociodemographic and clinical factors are expected to be related with the level of efficacy of the computerized multi-modal cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8-12 years.
* Manual Abilities Classification scale (MACs) ranging from I to III.
* An intelligible yes/no response system.
* Being able to understand simple instructions.
* Having the possibility of participating in the investigation for one year.
* Being able to access to internet at home.

Exclusion Criteria:

* Identified hearing or visual impairment that precludes neuropsychological assessment and training.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Spatial Span, Wechsler Nonverbal Scale of Ability (WNV)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Digit Span, Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Five Digit Test (FDT)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Auditory attention and Response Set, A Developmental NEuroPSYchological Assesment-II (NEPSY-II)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Word Generation, A Developmental NEuroPSYchological Assesment-II (NEPSY-II)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Tower Test, Delis-Kaplan Executive Function System (D-KEFS)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Conners' Continuous Performance Test-II (CPT-II)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Theory of Mind, A Developmental NEuroPSYchological Assesment-II (NEPSY-II)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Affect Recognition, A Developmental NEuroPSYchological Assesment-II (NEPSY-II)
Change from baseline Executive Function | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2)

SECONDARY OUTCOMES:
Change from baseline Visuoperception | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Benton Facial Recognition Test (BFRT)
Change from baseline Visuoperception | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Arrows, A Developmental NEuroPSYchological Assesment-II (NEPSY-II)
Change from baseline Memory | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Memory for designs, A Developmental NEuroPSYchological Assesment-II (NEPSY-II)
Change from baseline Memory | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Word selective reminding, Test of Memory and Learning (TOMAL)
Change from baseline Participation | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Participation and Environment Measure for Children and Youth (PEM-CY)
Change from baseline Quality of Life | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Cerebral Palsy Quality of Life (CP QOL-CHILD) questionnaire. CP QOL-CHILD is a proxy-reported questionnaire and QOL is measured as an index score (range from 0 to 100).
Change from baseline Structural and Functional neuroimaging | T0: 1 week before beginning; T1: 1 week immediately after training; T2: follow up (nine month after finished training)
  Structural and functional (resting state) magnetic resonance images (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Roser Pueyo, PhD, Principal Investigator — University of Barcelona
Locations (1):
- Facultat de Psicologia (Universitat de Barcelona), Barcelona, Spain

REFERENCES:
- [Derived] Garcia-Galant M, Blasco M, Moral-Salicru P, Soldevilla J, Ballester-Plane J, Laporta-Hoyos O, Caldu X, Miralbell J, Alonso X, Toro-Tamargo E, Melendez-Plumed M, Gimeno F, Leiva D, Boyd RN, Pueyo R. Understanding social cognition in children with cerebral palsy: exploring the relationship with executive functions and the intervention outcomes in a randomized controlled trial. Eur J Pediatr. 2024 Sep;183(9):3997-4008. doi: 10.1007/s00431-024-05635-y. Epub 2024 Jun 29. PMID 38951253
- [Derived] Garcia-Galant M, Blasco M, Laporta-Hoyos O, Berenguer-Gonzalez A, Moral-Salicru P, Ballester-Plane J, Caldu X, Miralbell J, Alonso X, Medina-Cantillo J, Povedano-Bullo E, Leiva D, Boyd RN, Pueyo R. A randomized controlled trial of a home-based computerized executive function intervention for children with cerebral palsy. Eur J Pediatr. 2023 Oct;182(10):4351-4363. doi: 10.1007/s00431-023-05072-3. Epub 2023 Jul 18. PMID 37462799
- [Derived] Garcia-Galant M, Blasco M, Reid L, Pannek K, Leiva D, Laporta-Hoyos O, Ballester-Plane J, Miralbell J, Caldu X, Alonso X, Toro-Tamargo E, Melendez-Plumed M, Gimeno F, Coronas M, Soro-Camats E, Boyd R, Pueyo R. Study protocol of a randomized controlled trial of home-based computerized executive function training for children with cerebral palsy. BMC Pediatr. 2020 Jan 7;20(1):9. doi: 10.1186/s12887-019-1904-x. PMID 31910803